CLINICAL TRIAL: NCT03276013
Title: Phase II Trial of Pembrolizumab in Combination With Doxorubicin in Advanced, Recurrent or Metastatic Endometrial Cancer (TOPIC)
Brief Title: Pembrolizumab in Combination With Doxorubicin in Advanced, Recurrent or Metastatic Endometrial Cancer
Acronym: TOPIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO17001
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Neoplasms
Keywords: Oncology; Endometrial Cancer; Pembrolizumab; Doxorubicin; Metastatic Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Non-randomized, single arm, multi-center, phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental): Doxorubicin 60 mg/kg IV over 30 minutes on day 1 every 3 weeks up to 9 cycles in combination with Pembrolizumab (MK-3475) 200 mg IV Q3W
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab in combination with doxorubicin

SUMMARY:
This is a non-randomized, single arm, multi-center, phase II study of pembrolizumab in combination with doxorubicin in subjects with recurrent/metastatic endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent/assent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research
2. Be >18 years of age on day of signing informed consent.
3. Have a histologically or cytologically-documented, advanced (metastatic and/or unresectable) endometrial carcinoma that is incurable and for which prior platinum-based chemotherapy for first-line treatment has failed. All epithelial endometrial histologies are eligible including: endometrioid, serous, clear-cell carcinoma, squamous or carcinosarcoma. Sarcomas and mesenchymal tumors are excluded.
4. Eligible subjects must have had only 1 prior line of systemic platinum-based chemotherapy for advanced, recurrent or metastatic endometrial cancer. Patients who have had 2 or more prior chemotherapeutic regimens for advanced, recurrent, or metastatic endometrial cancer are not allowed.

   Note: Prior neoadjuvant or adjuvant chemotherapy included in initial treatment may not be considered first- or later-line treatment unless such treatments were completed less than 6 months prior to the current tumor recurrence. Prior treatment may include chemotherapy, chemotherapy/radiation therapy, and/or consolidation/maintenance therapy.

   Prior hormonal treatment is not considered a line of therapy in any setting. Prior targeted therapy no directed against PD-1, PD-L1, PD-L2 pathway or any other immunemodulating mAb (including ipilimumab and any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) are allowed.
5. Have measurable disease based on RECIST 1.1, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm in long axis when measured by CT, MRI, or caliper measurement by clinical exam. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI. Tumor lesions situated in a previously irradiated area are considered measurable if progression according to RECIST 1.1 criteria has been demonstrated in such lesions. Patients must have radiographic evidence of disease progression following the most recent line of treatment. Areas of previous radiation may not serve as measurable disease unless there is evidence of progression post radiation according to RECIST 1.1 criteria. Patients with only one area of measureable disease that consent to have it biopsied are still eligible.
6. Availability of fresh or archival FFPE tumor specimens for analysis for biomarker analysis from a tumor lesion not previously irradiated (exceptions may be considered after Sponsor consultation). (See Procedure Manual for detailed instructions). Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion if archival specimen is not available. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 2, all screening labs should be performed within 7 days of treatment initiation.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential (Section 5.7.3) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Receipt of 2 or more prior chemotherapy regimens for advanced, recurrent, or metastatic endometrial cancer
3. History of myocardial infarction, acute inflammatory heart disease, unstable angina, or uncontrolled arrhythmia within the past 6 months.
4. Impaired cardiac function defined as left ventricular ejection fraction (LVEF) < 50 % (or below the study site's lower limit of normal) as measured by MUGA or ECHO. Planned concomitant use of potentially cardiotoxic medication.
5. Previous anthracycline-based chemotherapy.
6. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Has a known history of active TB (Bacillus Tuberculosis)
8. Hypersensitivity to pembrolizumab, doxorubicin or any of its excipients.
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Note: Palliative radiotherapy within 2 weeks prior to study is allowed provided that the site being treated is not subsequently used as a target lesions as per RECIST v.1.1 for the purpose of assessing tumor response on trial.
11. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
19. Has previously participated in any other pembrolizumab (MK-3475) trial, or received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or any other immunemodulating mAb (including ipilimumab and any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
20. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority. Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] Note: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.
21. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
22. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, social/ psychological issues.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
PFS rate at 6 months according to RECIST 1.1 criteria | 6 months
  To evaluate the efficacy of anti-PD1 blockade with pembrolizumab in combination with immunogenic chemotherapy with doxorubicin in patients with recurrent endometrial cancer in terms of patients who survived progression free (PFS) at least 6 months.

SECONDARY OUTCOMES:
To determine PFS rate at 6 months according to RECIST 1.1 criteria in the different groups by the genomic-The Cancer Genome Atlas (TCGA) classification; namely POLE, MSI, and Microsatellite Stable (MSS) | 6 months
To determine median PFS and ORR according to RECIST 1.1 criteria. | Through study completion, an average of 3 years
  PFS, defined as the time from allocation to the first documented disease progression according to RECIST 1.1 or death due to any cause, whichever occurs first. ORR will be used as the primary endpoint per RECIST 1.1 criteria, as assessed by investigators.
To determine median PFS and ORR according to RECIST 1.1 criteria in different genomic-TCGA subgroups | Through study completion, an average of 3 years
To determine median OS and OS rate | At 1, and 2-years
To evaluate median OS and OS rate at 1, and 2-years according to genomic-TCGA classification. | Through study completion, an average of 3 years
To evaluate DoR, defined as the time from first documented evidence of complete response (CR)or partial response (PR) until disease progression or death due to any cause, whichever occurs first | Through study completion, an average of 3 years
Number and grade of AEs, ECIs, SAEs, fatal SAEs, and laboratory changes that are Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Institut Català d'Oncologia L'Hospitalet (ICO L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía- Córdoba, Córdoba
  - CUN - Madrid, Madrid
  - El Centro Integral Oncológico Clara Campal (HM CIOCC),, Madrid
  - Hospital Universitario La Paz Madrid, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided